CLINICAL TRIAL: NCT05729776
Title: Comparison of the Glucose Metrics After Eating Pizza Margherita and a Meal Equivalent in Macronutrient in Pediatric Patients With Type 1 Diabetes Mellitus Treated With Hybrid Closed Loop Systems
Brief Title: Evaluation of the Glucose Metrics After Eating Pizza Margherita in Hybrid Closed Loop Users
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Angela Zanfardino, medical doctor, University of Campania Luigi Vanvitelli
Other Study IDs: PZ_2022
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Type1diabetes
Keywords: Glucose metrics; Pizza; Hybrid closed loop systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Overall eating pizza: All the patients that ate pizza
- Overall eating control meal: All patients that ate control mail (bread)
- Tandem patients eating pizza: All patients that ate pizza using Tandem Tslim system
- Medtronic 780 patients eating pizza: All patients that ate pizza using Medtronic 780 System

SUMMARY:
In previous study the investigators proved that blood glucose after eating pizza margherita could be managed with a simple wave bolus of insulin in pediatric patients with type 1 diabetes under controlled conditions. Participants in this previous study were Predictive Low Glucose Suspended (PLGS) System users. In this study the investigators want to demonstrate that blood glucose after the meal pizza margherita could also be managed with simple wave bolus of insulin in real life. The investigators will include just the patients with Hybrid Closed Loop (HCL) System.

DETAILED DESCRIPTION:
The investigators will enroll all patients with type 1 diabetes using of Hybrid Closed Loop (HCL) Systems (Medtronic MiniMed 780 G insulin pump system, Tandem T: Slim X2 insulin pump) followed in a diabetes center. The patients aged between 8- 18 will be included in the study just in a condition of using HCL Systems at least 3 months. Patients with HbA1c >8.5 % (69 mmol/mol), celiac disease, other food allergies will be excluded. The investigators will ask to parents feeding children with a pizza margherita which contains 100 grams of carbohydrates. Even if the patients could choose to consume pizza in different restaurants, the investigators will suggest having the pizza prepared with 200 grams of dough (which contains about 100 grams of carbohydrate). To validate the results the investigators will compare, for each patient, the data of glucose sensor and insulin pump after pizza consumption with those resulting from the consumption of a meal with the same macronutrient content. Patients should not consume anything else for 12 hours after the pizza (and after the meal containing the same macronutrient content). For this reason, patients will be encouraged to have these meals for dinner.

The aim of the study is comparing pizza with another meal which contains similar macronutrients. Second goal of this study is evaluating the blood glucose profile after eating pizza comparing the competency of two different Hybrid Closed Loop (HCL) Systems (Medtronic MiniMed 780 G insulin pump system, Tandem T: Slim X2 insulin pump) to manage blood glucose after eating pizza.

The investigators will collect data from both Carelink (for Medtronic device) and from Diasend (from Tandem device). All data will be exported in an excel file.

Demographic and clinical characteristic of enrolled patients (sex, BMI, Zscore BMI), HbA1c) will be collected from their medical records.

Observation period: from the dinner bolus to the next 10 hours of fasting.

Data from glucose sensor:

Endpoints from the sensor data will be evaluated:

* Percentage of time in targets with sensor glucose (SG) cut-offs of <54 mg/dl, ≤54>70mg/dl, ≥70<140mg/dl, ≥70 <180; ≥180<250 mg/dl and ≥250 mg/dl
* Coefficient of variation (%)
* Average Sensor Glucose SD (mg/dl) Times in target will be evaluated over the entire observation period (10 hours after bolus), from the bolus administration to 2 hours after administration, and from 2 to 5 hours after administration.

Data about insulin dose:

Endpoints from insulin pump will be evaluated:

* Total insulin dose (IU): it will be calculated as the sum of total basal insulin (IU) and total bolus insulin (IU) infused during the entire observation period.
* Total bolus amount (IU and %)
* Autocorrection bolus amount (IU and %)
* Autobasal amount (IU and %)

Data about carbohydrates amount:

Total carbohydrates amount entered during the observation period

Data about automatic mode:

Percentage of time in AutoMode during the observation period

The investigators will compare data of:

* "Pizza consumption" vs "control meal";
* "Medtronic pizza management" vs "Tandem T slim pizza management"

ELIGIBILITY:
Inclusion Criteria:

* The patients aged between 8- 18 will be included in the study just in a condition of using HCL Systems at least 3 months

Exclusion Criteria:

* Patients with HbA1c >8.5 % (69 mmol/mol), celiac disease, other food allergies will be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will enroll all patients with type 1 diabetes using of Hybrid Closed Loop (HCL) Systems (Medtronic MiniMed 780 G insulin pump system, Tandem T: Slim X2 insulin pump) followed in our diabetes center.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) after the consumption of pizza meal vs control meal | 10 hours
  TIR (Time in range:amount of time those with diabetes spend with blood glucose levels between 70 and 180 mg/dl)
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) after the consumption of pizza meal vs control meal | 10 hours
  TBR (Time below range:amount of time those with diabetes spend with blood glucose levels < 70 mg/dl)
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) after the consumption of pizza meal vs control meal | 10 hours
  TAR (Time Above Range: amount of time those with diabetes spend with blood glucose levels >250 mg/dl)

SECONDARY OUTCOMES:
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) in "Medtronic pizza management" and in "Tandem T slim pizza management" | 10 hours
  TIR (Time in range:amount of time those with diabetes spend with blood glucose levels between 70 and 180 mg/dl)
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) after "Medtronic pizza management" and"Tandem T slim pizza management" | 10 hours
  TBR (Time below range:amount of time those with diabetes spend with blood glucose levels < 70 mg/dl)
TIR, TBR and TAR evaluation(glucose metrics by glucose sensor) after "Medtronic pizza management" and"Tandem T slim pizza management" | 10 hours
  TAR (Time Above Range: amount of time those with diabetes spend with blood glucose levels >250 mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania, Naples, Italy

REFERENCES:
- [Result] Zanfardino A, Confetto S, Curto S, Cocca A, Rollato AS, Zanfardino F, Troise AD, Testa V, Bologna O, Stanco M, Piscopo A, Cohen O, Miraglia Del Giudice E, Vitaglione P, Iafusco D. Demystifying the Pizza Bolus: The Effect of Dough Fermentation on Glycemic Response-A Sensor-Augmented Pump Intervention Trial in Children with Type 1 Diabetes Mellitus. Diabetes Technol Ther. 2019 Dec;21(12):721-726. doi: 10.1089/dia.2019.0191. Epub 2019 Aug 8. PMID 31335171
- [Result] Della-Corte T, Gentile S, Di Blasi V, Guarino G, Corigliano M, Cozzolino G, Fasolino A, Martino C, Improta MR, Oliva D, Lamberti C, Vecchiato A, Vaia S, Satta E, Romano C, Alfarone C, Strollo F; Nefrocenter & Nyx Start-Up Research Study Group. Is pizza sutable to type 1 diabetes? A real life identification of best compromise between taste and low glycemic index in patients on insulin pump. Diabetes Metab Syndr. 2020 May-Jun;14(3):225-227. doi: 10.1016/j.dsx.2020.03.003. Epub 2020 Mar 12. PMID 32240944
- [Result] De Palma A, Giani E, Iafusco D, Bosetti A, Macedoni M, Gazzarri A, Spiri D, Scaramuzza AE, Zuccotti GV. Lowering postprandial glycemia in children with type 1 diabetes after Italian pizza "margherita" (TyBoDi2 Study). Diabetes Technol Ther. 2011 Apr;13(4):483-7. doi: 10.1089/dia.2010.0163. Epub 2011 Feb 28. PMID 21355715
- [Derived] Zanfardino A, Ippolito G, Ozen G, Galderisi A, Rollato AS, Chianese A, Testa V, Miraglia Del Giudice E, Scaramuzza AE, Iafusco D. Real-Life Performance of Automated Insulin Delivery Systems for High-Carbohydrate Meals: Are All Systems the Same? Diabetes Technol Ther. 2025 Aug;27(8):669-673. doi: 10.1089/dia.2025.0106. Epub 2025 Apr 2. PMID 40170658